CLINICAL TRIAL: NCT06998069
Title: Head and Neck Cancer Study Project in the Geriatric Population
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: The Miriam Hospital (Other); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 435
Record Dates: First submitted 2025-05-07; First posted 2025-05-31 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Neoplasms
Keywords: Squamous cell carcinoma of the head and neck; Geriatric population
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel; pembrolizumab; Radiotherapy; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I PD-L1 CPS 1-19 % (Other)
  Interventions: Drug: Arm I Carboplatin, Paclitaxel, Pembrolizumab
- Arm II PD-L1 CPS 0 (Other)
  Interventions: Drug: Arm II Carboplatin, Paclitaxel, Cetuximab
- Arm III PD-L1 CPS > or = 20% (Other)
  Interventions: Drug: Arm III Pembrolizumab

INTERVENTIONS:
Drug: Arm I Carboplatin, Paclitaxel, Pembrolizumab — Carboplatin, AUC 5, day 1 of each cycle, each cycle every 21 days for 4 cycles Paclitaxel, 175 mg/m2, day 1 of each cycle, each cycle every 21 days for 4 cycles Pembrolizumab, 200 mg, day 1 of each cycle, each cycle every 21 days for 4 cycles Radiation Therapy 30Gy 1 week
  Other Names: Radiation Therapy
  Arms: Arm I PD-L1 CPS 1-19 %
Drug: Arm II Carboplatin, Paclitaxel, Cetuximab — Carboplatin, AUC 5, day 1 of each cycle, each cycle every 21 days for 4 cycles Paclitaxel, 175 mg/m2, day 1 of each cycle, each cycle every 21 days for 4 cycles Cetuximab 400 mg/m2, day 1 of the first cycle and then 250 mg/m2 days 1, 8, 15 every 21 days for 4 cycles Radiation Therapy 30Gy 1 week
  Other Names: Radiation Therapy
  Arms: Arm II PD-L1 CPS 0
Drug: Arm III Pembrolizumab — Pembrolizumab, 200 mg, day 1 of each cycle, each cycle every 21 days for 4 cycles Radiation Therapy 30Gy 1 week
  Other Names: Radiation Therapy
  Arms: Arm III PD-L1 CPS > or = 20%

SUMMARY:
This is a study conducted in patients with a diagnosis of stage IB-IVA squamous cell carcinoma of the head and neck. Patients will have a comprehensive geriatric assessment (CGA) as part of standard assessments. The patients classified as frail, with a CGA score of 3-5, will then be treated with a novel reduced intensity regimen. The regimen will be tailored based on the programmed cell death ligand 1 combined positive score (PD-L1 CPS) and will involve 4 cycles of systemic chemotherapy and/or immunotherapy followed by radiation treatment.

DETAILED DESCRIPTION:
See above summary.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the following
* Pathology confirmed squamous cell carcinoma of the head and neck (unknown primary is excluded).
* Confirmed stage of disease between IB and IVA, based on imaging studies.
* CGA score of 3-5
* Evaluation by medical oncology and radiation oncology.
* Patients in the experimental group must be eligible for systemic treatment with chemoimmunotherapy followed by radiation treatment as determined by the geriatric oncology team.
* Age ≥ 65 years.
* ECOG performance status ≤ 2
* Adequate organ and marrow function as defined below:

Absolute neutrophil count ≥1.0 x 109/L Platelets >100,000/mm3 Total bilirubin <1.5 x ULN Aspartate aminotransferase (ast/sgot) <3 x ULN Alanine aminotransferase (alt/sgpt) <3 x ULN Creatinine clearance ≥ 40 mL/min as determined by Cockcroft Gault (using actual body weight) or <1.5 x Upper limit of normal

Males:

CLcr (mL/min) = "[140 - age (years)] × weight (kg)" /"72 × serum creatinine (mg/dL)"

Females:

(CLcr (mL/min) = "[140 - age (years)] × weight (kg)" /"72 × serum creatinine (mg/dL)" × 0.85

* Patients receiving pembrolizumab must meet standard institutional criteria for immunotherapy including no history of severe autoimmune disease.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with metastases, including treated brain metastases, are not eligible for enrollment.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have previously received systemic chemoimmunotherapy for H/N cancer.
* Patients with uncontrolled intercurrent illness.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Completion | Approximately 14 weeks
  Number of participants who complete 4 cycles of systemic therapy followed by one week of radiation therapy within 14 weeks from start of therapy

SECONDARY OUTCOMES:
Assessment of the Overall Response Rate (ORR). | Approximately 12 weeks after completion of the treatment
  Number of participants who achieve a complete or partial response rate per RECIST criteria
Assessment of the Disease-Free Survival (DFS) and Overall Survival (OS). | Approximately 3 years
  Number of participants who have no evidence of disease and/or who are alive
Toxicity Assessment | Approximately 30 days post treatment
  Participants toxicity assessment (side effects) will be graded per the National Cancer Institute's (NCI) common terminology criteria for adverse events (CTCAE v5.0) reporting.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island and The Miriam Hospitals, Providence, Rhode Island, United States